CLINICAL TRIAL: NCT04529174
Title: Evaluation of an Oral Nutritional Supplement for Effect on Total High-Density Lipoprotein (HDL) Cholesterol, HDL Functionality, Particle Size and Number
Brief Title: Oral Nutritional Supplement Effect on HDL Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metagenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HTI-003
Record Dates: First submitted 2020-08-21; First posted 2020-08-27 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: HDL
Keywords: HDL cholesterol; HDL function; HDL particle; Dietary supplement; Nutraceutical
MeSH Terms: conditions — Huntington Disease-Like 2

STUDY DESIGN:
Intervention Model Description: Randomized double-blind Placebo controlled trial. Dietary
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active HDL supplement (Active Comparator): 25 subjects (ages 18-85 years old) will receive an active HDL supplement (CardioLux™HDL). They will take 2 capsules twice a day with food for 12 weeks. Total daily dosing is four (4) capsules.
  Interventions: Dietary Supplement: CardioLux™HDL
- Placebo (Placebo Comparator): 25 randomly selected subjects (ages 18-85 years old) will receive a matching Placebo. They will take 2 capsules twice each day with food for 12 weeks. Total daily dosing is four (4) capsules.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CardioLux™HDL — Enrollment will occur according to the inclusion/ exclusion criteria and after the review and signing of the Informed Consent form. Clinical testing will be performed at baseline and each visit (2, 3).
  Measurement of height, weight with body composition analysis, body mass index, waist circumference, and vital signs (blood pressure, heart rate) will be measured.
  Review of medical history and current medications by clinician; and collection of fasting blood for testing of the complete blood count (CBC), comprehensive metabolic profile (CMP), as well as a urine pregnancy test in females of child-bearing potential.
  Visits: Baseline (Visit 1), Week 6 (Visit 2) and Week 12 (Visit 3/End of Study)
  Arms: Active HDL supplement
Dietary Supplement: Placebo — Enrollment will occur according to inclusion /exclusion criteria and after the review and signing of the Informed Consent form. Clinical testing will be performed at baseline and each visit (2, 3).
  Measurement of height, weight with body composition analysis, body mass index, waist circumference, and vital signs (blood pressure, heart rate) will be measured.
  Review of medical history and current medications by clinician; and collection of fasting blood for testing of the complete blood count (CBC), comprehensive metabolic profile (CMP), as well as a urine pregnancy test in females of child-bearing potential.
  Visits: Baseline (Visit 1), Week 6 (Visit 2) and Week 12 (Visit 3/End of Study)
  Arms: Placebo

SUMMARY:
Evaluate the effects of a proprietary supplement on total HDL, HDL functionality, HDL particle size and HDL particle number (HDL-P)

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female patients or female patients of childbearing age on contraception age 18-80years.
* Total HDL level 38mg/dL or lower in men and HDL 45 mg/dL or lower in women and a low HDL-P defined as less than 7000 by Spectracell LPP Plus.
* CHL HDL Fx score equal to or greater than 0.9.
* Patients will remain on their present diet, exercise program, medications (except for those who alter serum lipids) sleeping habits, alcohol intake, caffeine intake, smoking amount and emotional status as best as possible related to stress and anxiety and maintain body weight at baseline visit as best as possible to avoid confounding variables.
* No other lipid lowering supplement can be taken during the study.
* All lipid lowering supplements must have been discontinued at least 30 days prior t o study entry.

Exclusion Criteria:

* Pregnant females
* Females of childbearing age not on an accepted contraception control method
* Previous myocardial infarction within 5 years
* Unstable angina
* Previous stroke or TIA within 5 years
* Uncompensated congestive heart failure
* Previous PCTA or stent within 5 years
* Previous CABG within 5 years
* Patients on statins, fibrates, or other lipid lowering medications or any supplement known to affect serum lipids.
* Known or previous cancer within 5 years
* Type 1 diabetes mellitus
* Kidney disease as defined by serum creatinine over 2.5 mg/dL

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
HDL-FX test HDL-FX test | Change from Baseline to End of Study (week 12)
  Reverse Cholesterol Transport (RCT)(CEC) with Cleveland Heart Lab (CHL)
HDL mapping | Change from Baselineto End of study (week 12)
  HDL mapping with Boston Heart Lab (BHL)

SECONDARY OUTCOMES:
Myloperoxidase (MPO) | Change from Baseline to End of Study (week 12)
  measured with Quest Lab test
LP-PLA-2 test | Change from Baseline to End of Study (week 12)
  Measured with Quest Lab test
Dietary Intake | Change from Baseline to End of Study (week 12)
  24 hour recall

OTHER OUTCOMES:
Weight | Change from Baseline to End of Study (week 12)
  measured in pounds (Lbs)
Body Mass Index | Change from Baseline to End of Study (week 12)
  measured in kg/m2
Waist Circumference | Change from Baseline to End of Study (week 12)
  measured in cm
Blood pressure (systolic/diastolic) | Change from Baseline to End of Study (week 12)
  measured in mm Hg

CONTACTS AND LOCATIONS:
Overall Officials: Mark Houston, MD, Principal Investigator — Hypertension Institute
Locations (1):
- Hypertension Institute, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No